CLINICAL TRIAL: NCT01289028
Title: An Open-label, Multi-center Study to Evaluate the Efficacy of Nilotinib in Adult Patients With Gastrointestinal Stromal Tumors Resistant to Imatinib and Sunitinib.
Brief Title: Efficacy of Nilotinib in Adult Patients With Gastrointestinal Stromal Tumors Resistant to Imatinib and Sunitinib.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CAMN107DDE05; 2008-000357-35 (EudraCT Number)
Record Dates: First submitted 2011-01-16; First posted 2011-02-03 (Estimated); Results first posted 2016-11-01 (Estimated); Last update posted 2017-01-02 (Estimated); Status verified 2016-06

CONDITIONS: Gastrointestinal Stromal Tumors
Keywords: GIST; Imatinib; Sunitinib; Gastrointestinal; Stromal; Tumors
MeSH Terms: conditions — Gastrointestinal Stromal Tumors; Neoplasms | interventions — nilotinib

ARMS (1):
- Nilotinib (Experimental): nilotinib 400 mg twice daily (bid).
  Interventions: Drug: Nilotinib

INTERVENTIONS:
Drug: Nilotinib
  Other Names: AMN107

SUMMARY:
This study will evaluate the preliminary efficacy of nilotinib in pretreated patients (Imatinib, Sunitinib) with unresectable or metastatic gastrointestinal stromal tumors.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed diagnosis of GIST that is unresectable and/or metastatic and therefore not amenable to surgery or combined modality with curative intent.
* Radiologically confirmed disease progression during imatinib therapy at a dose of at least 400 mg daily and/or radiologically confirmed disease progression during sunitinib therapy OR documented intolerance to imatinib and/or sunitinib. (Patients with prior additional investigational treatment of GIST prior to study entry can be included.)
* At least one measurable site of disease on CT/MRI as defined by RECIST criteria.

Exclusion Criteria:

* Prior treatment with nilotinib.
* Treatment with any cytotoxic and/or investigational cytotoxic drug ≤ 4 weeks (6 weeks for nitrosurea or mitomycin C) prior to Visit 1.
* Prior or concomitant malignancies requiring active treatment other than GIST with the exception of previous or concomitant basal cell skin cancer, previous cervical carcinoma in situ.
* Impaired cardiac function at visit 1
* Patients with severe and/or uncontrolled concurrent medical disease that in the opinion of the investigator could cause unacceptable safety risks or compromise compliance with the protocol e.g. impairment of gastrointestinal (GI) function, or GI disease that may significantly alter the absorption of the study drugs, uncontrolled diabetes.

Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 125 (Actual)
Dates: Start 2008-11; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (18):
- Germany (11):
  - Novartis Investigative Site, Bad Saarow
  - Novartis Investigative Site, Dresden
  - Novartis Investigative Site, Düsseldorf
  - Novartis Investigative Site, Essen
  - Novartis Investigative Site, Frankfurt
  - Novartis Investigative Site, Freiburg im Breisgau
  - Novartis Investigative Site, Halle
  - Novartis Investigative Site, Hanover
  - Novartis Investigative Site, Mannheim
  - Novartis Investigative Site, München
  - Novartis Investigative Site, Ulm
- Italy (7):
  - Novartis Investigative Site, Bologna, BO
  - Novartis Investigative Site, Genova, GE
  - Novartis Investigative Site, Taormina, ME
  - Novartis Investigative Site, Milan, MI
  - Novartis Investigative Site, Padua, PD
  - Novartis Investigative Site, Aviano, PN
  - Novartis Investigative Site, Torino, TO

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Nilotinib
Started | 125
Completed | 42
Not Completed | 83
Not completed — Progressive Disease | 49
Not completed — Adverse Event | 14
Not completed — Withdrawal by Subject | 6
Not completed — Death | 4
Not completed — Lack of Efficacy | 2
Not completed — No longer required | 2
Not completed — Lost to Follow-up | 2
Not completed — New Cancer Therapy | 2
Not completed — Abnormal Lab Value | 1
Not completed — Missing reason for discon | 1

BASELINE CHARACTERISTICS:
Arm/Group | Nilotinib
Number analyzed (Participants) | 125
Age, Continuous [Mean (Standard Deviation); unit: years] | 60 (12.1)
Gender [Count of Participants; unit: Participants]
  Female | 46
  Male | 79

OUTCOME MEASURES:

1. Primary Outcome: Percent of Patients Achieving Stable Disease (SD)
Description: Neither sufficient shrinkage to qualify for Partial Response nor sufficient increase to qualify for Progression Disease, taking as reference the smallest sum of the longest diameter since the treatment started.
Time Frame: During the first 4 months
Measure: Number; unit: % participants
Arm/Group | Nilotinib
Number analyzed (Participants) | 125
% participants | 48.8

2. Primary Outcome: Percent of Patients Achieving Partial Response (PR)
Description: The primary efficacy variable was defined as the proportion of patients with a best overall response of CR by Week 16/Month 4 based on local assessment according to RECIST (Version 1.0). This is an at least a 30% decrease in the sum of the longest diameter of target lesions, taking as reference the baseline sum longest diameter.
Time Frame: during the first 4 months
Population: ITT set, N=125
Measure: Number; unit: percentage of participants
Arm/Group | Nilotinib
Number analyzed (Participants) | 125
percentage of participants | 0

3. Primary Outcome: Percent of Patients Achieving Complete Response (CR)
Description: Complete response (CR) is the Disappearance of all target lesions.
Time Frame: during the first 4 months
Measure: Number; unit: percentage of participants
Arm/Group | Nilotinib
Number analyzed (Participants) | 125
percentage of participants | 0

4. Secondary Outcome: Analysis of Time to Overall Response (CR or PR) According to RECIST Using Kaplan-Meier Method for ITT Population
Description: Complete Response (CR): Disappearance of all target lesions. and Partial Response (PR): At least a 30% decrease in the sum of the longest diameter of target lesions, taking as reference the baseline sum longest diameter.
Time Frame: 24 weeks and 52 weeks
Population: ITT population
Measure: Number; unit: percentage of participants
Groups:
- Nilotinib: ITT
Arm/Group | Nilotinib
Number analyzed (Participants) | 125
percentage of participants
  24 weeks | 92.0
  52 weeks | 92.0

5. Secondary Outcome: Time to Overall Response (CR or PR): Per Protocol Population
Description: Complete Response (CR): Disappearance of all target lesions, and Partial Response (PR): At least a 30% decrease in the sum of the longest diameter of target lesions, taking as reference the baseline sum longest diameter.
Time Frame: 24 weeks and 52 weeks
Measure: Number; unit: percentage of participants
Groups:
- Nilotinib: Per Protocol population
Arm/Group | Nilotinib
Number analyzed (Participants) | 98
percentage of participants
  24 weeks | 91.2
  52 weeks | 91.2

6. Secondary Outcome: Time to Tumor Progression
Description: Time to tumor progression defined as the time from start of treatment to observed tumor progression (censoring for death without progression) as stated in the original protocol was not evaluated as stated in section 9.8.3 of the clinical study report.
Time Frame: during the first 4 months
Population: Time to tumor progression defined as the time from start of treatment to observed tumor progression (censoring for death without progression) as stated in the original protocol was not evaluated
Arm/Group | Nilotinib
Number analyzed (Participants) | 0

7. Secondary Outcome: Duration of Overall Response
Description: The best overall response is the best response recorded from the start of the treatment until disease progression/recurrence
Time Frame: during 12 months
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Nilotinib
Number analyzed (Participants) | 125
days | 1331 [366 to NA] — Due to number of censored cases (insufficient number of participants with measurable events) Upper Limit CI was not possible to calculate.

8. Secondary Outcome: Overall Survival, Number of Events Related to Progression of the Disease
Description: The OS rate could not be calculated due to the high number of censored cases. Number of censored, n (%) 108 (86.4). Only available data is number of events. OS was defined as the time from first study drug administration to death from any cause. If a patient was not known to have died, survival was censored at date of last contact.
Time Frame: during 12 months
Measure: Number; unit: events
Arm/Group | Nilotinib
Number analyzed (Participants) | 125
events | 17

9. Secondary Outcome: Progression Free Survival (PFS) of the Patients Who Were Included Due to an Intolerability of a Prior Treatment.
Description: Progression-free survival (PFS) is defined as the time from first study drug administration to objective tumor progression or death from any cause. If a patient has not had an event, PFS is censored at the date of last adequate tumor assessment.
Time Frame: during 12 months
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Nilotinib
Number analyzed (Participants) | 125
days | 110 [64 to 118]

ADVERSE EVENTS:
Groups:
- All Patients: All patients
Arm/Group | All Patients
Serious Adverse Events (participants affected / at risk) | 60/125
Other Adverse Events (participants affected / at risk) | 107/125
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | All Patients (N=125)
Anaemia (Blood and lymphatic system disorders) | 6
Acute coronary syndrome (Cardiac disorders) | 1
Angina unstable (Cardiac disorders) | 1
Aortic valve stenosis (Cardiac disorders) | 1
Atrial fibrillation (Cardiac disorders) | 1
Cardiac failure (Cardiac disorders) | 1
Coronary artery stenosis (Cardiac disorders) | 1
Myocardial infarction (Cardiac disorders) | 2
Abdominal pain (Gastrointestinal disorders) | 7
Abdominal pain upper (Gastrointestinal disorders) | 1
Abdominal wall mass (Gastrointestinal disorders) | 1
Ascites (Gastrointestinal disorders) | 2
Constipation (Gastrointestinal disorders) | 3
Diarrhoea (Gastrointestinal disorders) | 1
Flatulence (Gastrointestinal disorders) | 1
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
Melaena (Gastrointestinal disorders) | 1
Mesenteric haemorrhage (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 2
Pancreatitis acute (Gastrointestinal disorders) | 1
Subileus (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 5
Asthenia (General disorders) | 1
Chest pain (General disorders) | 1
Chills (General disorders) | 1
Condition aggravated (General disorders) | 2
Device occlusion (General disorders) | 2
Disease progression (General disorders) | 6
Fatigue (General disorders) | 3
General physical health deterioration (General disorders) | 3
Multi-organ failure (General disorders) | 1
Obstruction (General disorders) | 1
Pyrexia (General disorders) | 5
Cholangitis (Hepatobiliary disorders) | 1
Cholestasis (Hepatobiliary disorders) | 1
Hepatotoxicity (Hepatobiliary disorders) | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 1
Breast abscess (Infections and infestations) | 1
Infected skin ulcer (Infections and infestations) | 1
Infection (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 1
Rectal abscess (Infections and infestations) | 1
Sinusitis (Infections and infestations) | 1
Staphylococcal infection (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 1
Alcohol poisoning (Injury, poisoning and procedural complications) | 1
Concussion (Injury, poisoning and procedural complications) | 1
Lip injury (Injury, poisoning and procedural complications) | 1
Amylase increased (Investigations) | 1
Blood creatinine increased (Investigations) | 2
C-reactive protein increased (Investigations) | 2
Electrocardiogram QT prolonged (Investigations) | 1
Gamma-glutamyltransferase increased (Investigations) | 1
Haemoglobin decreased (Investigations) | 1
Lipase increased (Investigations) | 2
Weight decreased (Investigations) | 2
Cachexia (Metabolism and nutrition disorders) | 1
Decreased appetite (Metabolism and nutrition disorders) | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 1
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3
Metastases to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3
Intercostal neuralgia (Nervous system disorders) | 1
Hydronephrosis (Renal and urinary disorders) | 1
Renal failure (Renal and urinary disorders) | 2
Renal failure acute (Renal and urinary disorders) | 1
Ureteric stenosis (Renal and urinary disorders) | 1
Urethral stenosis (Renal and urinary disorders) | 1
Urinary retention (Renal and urinary disorders) | 1
Urinary tract obstruction (Renal and urinary disorders) | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1
Arterial occlusive disease (Vascular disorders) | 1
Peripheral arterial occlusive disease (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | All Patients (N=125)
Anaemia (Blood and lymphatic system disorders) | 14
Abdominal pain (Gastrointestinal disorders) | 28
Abdominal pain upper (Gastrointestinal disorders) | 7
Constipation (Gastrointestinal disorders) | 32
Diarrhoea (Gastrointestinal disorders) | 18
Flatulence (Gastrointestinal disorders) | 13
Nausea (Gastrointestinal disorders) | 28
Vomiting (Gastrointestinal disorders) | 21
Asthenia (General disorders) | 10
Fatigue (General disorders) | 44
Oedema peripheral (General disorders) | 17
Pyrexia (General disorders) | 19
Nasopharyngitis (Infections and infestations) | 12
Alanine aminotransferase increased (Investigations) | 8
Blood alkaline phosphatase increased (Investigations) | 16
C-reactive protein increased (Investigations) | 9
Lipase increased (Investigations) | 7
Transaminases increased (Investigations) | 7
Weight decreased (Investigations) | 14
Decreased appetite (Metabolism and nutrition disorders) | 18
Hypophosphataemia (Metabolism and nutrition disorders) | 7
Arthralgia (Musculoskeletal and connective tissue disorders) | 8
Back pain (Musculoskeletal and connective tissue disorders) | 11
Muscle spasms (Musculoskeletal and connective tissue disorders) | 9
Myalgia (Musculoskeletal and connective tissue disorders) | 10
Pain in extremity (Musculoskeletal and connective tissue disorders) | 11
Headache (Nervous system disorders) | 14
Cough (Respiratory, thoracic and mediastinal disorders) | 8
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 8
Alopecia (Skin and subcutaneous tissue disorders) | 10
Dry skin (Skin and subcutaneous tissue disorders) | 10
Pruritus (Skin and subcutaneous tissue disorders) | 21
Rash (Skin and subcutaneous tissue disorders) | 10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.